CLINICAL TRIAL: NCT04406896
Title: An Open-label, Single-dose, Phase 1 Study to Evaluate the Pharmacokinetics of Selatogrel in Subjects With Mild and Moderate Hepatic Impairment Compared to Matched Healthy Subjects
Brief Title: The Effect of Reduced Liver Function on Selatogrel Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viatris Innovation GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ID-076-108; 2020-001315-25 (EudraCT Number)
Record Dates: First submitted 2020-05-25; First posted 2020-05-29 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2022-11

CONDITIONS: Healthy Subjects; Hepatic Impairment
MeSH Terms: interventions — selatogrel

STUDY DESIGN:
Intervention Model Description: Moderate hepatic impaired participants will be dosed after an interim analysis of at least 6 participants with mild hepatic impairment. Healthy participants will be matched to hepatic impaired participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Participants with mild hepatic impairment (Group 1) (Experimental): Participant with Child-Pugh Grade A Score of 5-6.
  Interventions: Drug: Selatogrel
- Participants with moderate hepatic impairment (Group 2) (Experimental): Participant with moderate hepatic impairment with a Child-Pugh Grade B Score of 7-9.
  Interventions: Drug: Selatogrel
- Healthy participants (Group 3) (Experimental)
  Interventions: Drug: Selatogrel

INTERVENTIONS:
Drug: Selatogrel — A single subcutaneous injection of 16 mg.
  Other Names: ACT-246475

SUMMARY:
This is a prospective, single-center, open-label, single-dose, Phase 1 study, to assess the effect of mild and moderate hepatic impairment due to liver cirrhosis on the pharmacokinetics of selatogrel (ACT-246475).

ELIGIBILITY:
Inclusion Criteria:

All participants (Groups 1,2 and 3)

* Signed informed consent in a language understandable to the participant prior to any study-mandated procedure.
* Male or female participant aged between 18 and 79 years (inclusive) at screening.
* Body mass index of 18.0 to 35.0 kg/m2 (inclusive) at screening.
* Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test on Day 1 (pre-dose). They must consistently and correctly use (from screening, during the entire study, and for at least 30 days after last study treatment administration) an acceptable effective method of contraception method, be sexually inactive, or have a vasectomized partner. If a hormonal contraceptive is used, it must have been initiated at least 1 month before treatment administration.
* Women of non-childbearing potential.

Additional principal inclusion criteria for participants with hepatic impairment (Groups 1 and 2)

* Hepatic impairment due to liver cirrhosis according to the Child-Pugh classification:

  * Group 1: Mild hepatic impairment, Child-Pugh A = score 5-6.
  * Group 2: Moderate hepatic impairment, Child-Pugh B = score 7-9.
* Systolic blood pressure (SBP) 95-160 mmHg, diastolic blood pressure (DBP) 60-95 mmHg, and pulse rate 50-100 bpm (inclusive), measured on the same arm, after 5 minutes in the supine position at screening and on Day 1 (pre-dose).
* Estimated glomerular filtration rate (eGFR) at screening using the Modification of Diet in Renal Disease (MDRD) formula of:

  * greater than or equal to 60 mL/min/1.73 m2 for participants with mild hepatic impairment (Group 1)
  * greater than or equal to 45 mL/min/1.73 m2 for participants with moderate hepatic impairment (Group 2).
* Stable concomitant medications for at least 3 weeks prior to screening and up to Day 1 and expected to be stable during the conduct of the study.

Additional principal inclusion criteria for healthy participants (Group 3)

* Normal blood pressure measured on the same arm, after 5 minutes in the supine position at screening and on Day 1 pre-dose defined as:

  * SBP 90 to 140 mmHg, DBP 60 to 90 mmHg, and pulse rate 50 to 100 bpm (inclusive) for participants less than 60 years of age.
  * SBP 95 to 160 mmHg, DBP 65 to 95 mmHg, and pulse rate 50 to 100 bpm (inclusive) for participants 60 years and older.
* eGFR greater than or equal to 80 mL/min/1.73 m2 at screening using the MDRD formula.

Exclusion Criteria:

All participants (Groups 1, 2 and 3)

* Pregnant or lactating woman.
* Previous exposure to selatogrel.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* Known hypersensitivity to P2Y12 receptor antagonists or any excipients of the drug formulation.
* Known platelet disorders.
* Legal incapacity or limited legal capacity at screening.

Additional exclusion criteria for participants with hepatic impairment (Groups 1 and 2)

* History or clinical evidence of any disease and/or existence of any surgical or medical condition (e.g., cholecystectomy), which might interfere with the absorption, distribution, metabolism, and excretion (ADME) of the study treatment (except for hepatic impairment, appendectomy, and herniotomy).
* Acute hepatitis, hepatic cancer, primary biliary cirrhosis, or any form of cholestatic disease.
* Clinical evidence or suspected acute liver failure as judged by the investigator.
* Severe ascites and/or pleural effusion.
* Encephalopathy greater than grade 2.
* Clinical evidence of current alcohol or drug abuse.
* Clinically relevant abnormalities on a 12-lead ECG, except for abnormalities related to hepatic impairment, after 5 minutes in the supine position at screening and on Day 1 pre-dose.

Additional exclusion criteria for healthy participants (Group 3)

* History or clinical evidence of any disease and/or existence of any surgical or medical condition (e.g., cholecystectomy), which might interfere with the ADME of the study treatment (except for appendectomy and herniotomy).
* History or clinical evidence of alcohol or drug abuse within the 3 years prior to screening.
* Family or personal history of prolonged bleeding or bleeding disorders, intracranial vascular diseases, stroke, reasonable suspicion of vascular malformations, or peptic ulcers.
* Previous treatment with any prescribed medications or over-the-counter medications within 2 weeks or 5 times the terminal half-life (t½), whichever is longer prior to study treatment administration (excludes contraceptives and hormone replacement therapy).

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) of selatogrel | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 3.
Time to reach Cmax (tmax) | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 3.
Area under the plasma concentration-time curves (AUC0-t) of selatogrel | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 3.
The area under the plasma concentration-time curve from zero to infinity (AUC0-inf) of selatogrel | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 3.
Terminal half-life (t½) of selatogrel | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 3.
The apparent clearance (CL/F) of selatogrel | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 3.
The apparent volume of distribution (Vz/F) of selatogrel | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose) up to Day 3.
Plasma protein binding of selatogrel | Multiple pharmacokinetic sampling at predefined times on Day 1 (pre-dose and post-dose).

SECONDARY OUTCOMES:
Change from baseline in supine blood pressure | Multiple predefined times on Day 1 (pre-dose) up to Day 3.
Change from baseline in temperature | Multiple predefined times on Day 1 (pre-dose) up to Day 3.
Change from baseline in pulse rate | Multiple predefined times on Day 1 (pre-dose) up to Day 3.
Change from baseline in body weight | Multiple predefined times on Day 1 (pre-dose) up to Day 3.
Change from baseline in clinical laboratory tests | Multiple predefined times on Day 1 (pre-dose) up to Day 3.
Change from baseline at each time point of measurement in ECG variables. | Multiple predefined times on Day 1 (pre-dose) up to Day 3.
Inhibition of platelet aggregation | Multiple predefined times on Day 1 (pre-dose) up to Day 3.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Viatris Innovation GmbH
Locations (1):
- CRS Clinical Research Services, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No